CLINICAL TRIAL: NCT05396352
Title: Cerebellum and Autism: Regional Specialization for Social and Executive Functions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Catherine Stoodley, Associate Professor, American University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: R15MH126404 (NIH); R15MH126404 (NIH)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Autism; Autism Spectrum Disorder
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Within-subjects design (active, sham tDCS) with separate groups receiving tDCS targeting cerebellar right lobule VII and the posterior cerebellar vermis.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Right cerebellum (Experimental): Participants (neurotypical, autistic) in this arm will receive tDCS targeting the right posterolateral cerebellum (lobule VII). All participants will receive anodal, cathodal and sham tDCS.
  Interventions: Device: Transcranial direct current stimulation
- Posterior vermis (Experimental): Participants (neurotypical, autistic) in this arm will receive tDCS targeting the posterior cerebellar vermis. All participants will receive anodal, cathodal and sham tDCS.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — TDCS involves applying small (1-2 mA) electric currents to the scalp in order to transiently modify local neuronal electrical potentials in the brain.
  Other Names: tDCS

SUMMARY:
The goal of this study is to determine the impact of neuromodulation to the cerebellum on social and executive functions in neurotypical young adults and young adults with autism.

DETAILED DESCRIPTION:
Autism spectrum disorder is a prevalent neurodevelopmental condition characterized by deficits in social communication and the presence of repetitive and inflexible behaviors. There are currently few biologically-targeted treatment options for autism, in part because the underlying neurobiology is not well understood. One region of the brain that is consistently implicated in autism is the cerebellum. Specifically, two cerebellar subregions show structural and functional differences in autism: right cerebellar lobule VII (RVII) and the posterior cerebellar vermis. Based on the different anatomical connectivity of these regions, the investigators hypothesize that RVII and the posterior vermis regulate different core deficits in autism. In this study, the investigators combine cerebellar neuromodulation with functional neuroimaging to test the hypothesis that neuromodulation targeting RVII will selectively alter social learning and neural networks supporting social behavior, while neuromodulation targeting the posterior vermis will impact cognitive flexibility and neural networks involved in the allocation of attention. Neurotypical adults and adults with autism will complete social and cognitive flexibility tasks after excitatory, inhibitory, or sham neuromodulation in a within-subjects design. Some participants will receive neuromodulation targeting RVII and others will receive neuromodulation targeting the posterior vermis. The investigators will acquire functional brain imaging data during and after cerebellar neuromodulation, which will allow the team to better understand the mechanisms by which non-invasive neuromodulation might impact behavior in clinical disorders.

ELIGIBILITY:
Please note: This study takes place at American University and Georgetown University in Washington, DC. We do not have funds for travel and lodging available for this study, so participants should be local to the DC region.

Inclusion Criteria:

All participants

* Aged 18-35
* Able to provide written, informed consent
* NIH Toolbox age-adjusted Cognitive Function Composite standard score ≥ 85
* Native English speaker
* Right-handed
* Not pregnant
* Able to attend all study sessions
* Pass safety screening for MRI and neuromodulation (e.g. no metal in body, implanted devices, history of seizure, claustrophobia)

Additional INCLUSION criteria for adults with autism Either

* Prior research-reliable diagnosis of autism spectrum disorder (ASD) Or
* Meet DSM-5 criteria for ASD confirmed with ADOS-2 via research-reliable clinical assessment

Exclusion Criteria:

Neurotypical adults

* Age <18 or >35
* NIH Toolbox age-adjusted Cognitive Function Composite standard score < 85
* Contraindications for MRI or neuromodulation with tDCS (e.g. metal in body, pacemaker or other implanted device, history of seizure, claustrophobia)
* Current or prior history of neurological or neurodevelopmental condition or brain injury
* Psychotropic medication
* Pregnancy

Adults with autism

* Age <18 or >35
* Participants with a legal authorized representative
* NIH Toolbox age-adjusted Cognitive Function Composite standard score < 85
* Contraindications for MRI or neuromodulation with tDCS (e.g. metal in body, pacemaker or other implanted device, history of seizure, claustrophobia)
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Reading the Mind in the Eyes Test Adult Version | Within 30min post-tDCS
Cyberball social ball-playing task | Within 30min post-tDCS
Flexible Item Selection Test | Within 30min post-tDCS
Functional MRI data | Within 45min post-tDCS
  Functional MRI task data and resting state functional connectivity data

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gunthert, Ph.D., Principal Investigator — American University
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data, including scores of behavioral tests and skull-stripped brain images, may be shared upon personal request after initial manuscripts based on this work have been published. Individuals wishing to use these data must agree not to attempt to identify participants or redistribute the data, to destroy the data after analyses are completed, and to acknowledge the data resource in any presentations or publications. For participants that consent to having their de-identified data shared with the National Database for Autism Research (NDAR), we will submit data to NDAR in accordance with the NIH guidelines (http://ndar.nih.gov/contribute.html).
Supporting Information: Study Protocol
Time Frame: Data uploaded to NDAR will be released following study completion
Access Criteria: * Access to NDAR
  * Individuals wishing to use these data must agree not to attempt to identify participants or redistribute the data, to destroy the data after analyses are completed, and to acknowledge the data resource in any presentations or publications.
URL: http://nda.nih.gov